CLINICAL TRIAL: NCT06853652
Title: Maintenance-phase PROtein Requirements After RouX-en-Y-gastric Bypass Surgery
Brief Title: Protein Requirements After Bariatric Surgery
Acronym: PROXY
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S69673
Record Dates: First submitted 2025-02-21; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Obesity and Overweight; Bariatric Surgery (Gastric Bypass); Protein Requirement
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Male adults with previous RYGB surgery: Male adults with previous RYGB surgery

SUMMARY:
The study investigates protein requirements at least 1 year after gastric bypass surgery in adult males, to investigate whether protein requirements are elevated compared to protein requiremens for the general populaiotn. The main study outcome is the estimated average protein requirements for the study populaiton.

DETAILED DESCRIPTION:
The study objective is to determine maintenance dietary protein requirements for adult males who have previously undergone Roux-en-Y-Bypass (RYGB) surgery, using the minimally invasive Indicator Amino Acid Oxidation (IAAO) method. The study hypothesis is that dietary protein requirements will be elevated in this population compared to young adults with no previous bariatric surgery. The null hypothesis states that there is no difference in dietary protein requirements between adults with previous RYGB surgery and adults without previous surgery. Protein requirements will be expressed relative to fat-free-mass (FFM) to account for obesity-related increases in lean mass.

The primary endpoint of the study is the estimated average protein requirements (g/kg FFM/d) and the upper limit of the 95% confidence interval.

The study comprises a nutritional experimental study using the IAAO method to determine protein requirements. Indicator amino acid oxidation is measured at seven incremental protein intake levels, each on a separate study day after two adaptation days. Protein intake requirements are calculated as the protein intake level where the indicator amino acid oxidation ceases to decline further despite a further increase in protein intake. This is referred to as the breakpoint. The sequences of protein intake levels are randomized for each study participant. Protein requirements are calculated, not per individual, but for the whole study population, when sufficient oxidation studies are included at each protein intake level. This implies that the same individual does not have to complete all the oxidation studies at the seven time points.

The study will consist of one initial screening and planning visit, and 2 to 7 metabolic trial visits. Each participant can complete at least two, preferably more, and up to all 7 protein intake levels.

Patients who previously consented to be included in a UZ Leuven Obesity Clinic repository (ClinicalTrials.gov Identifier NCT04614961; S-62590) will be pre-screened according to the study criteria. Thereafter patients who remain eligible will be contacted and will receive information regarding the study using the informed consent form. An invitation to participate in the study will also be circulated through patient support groups of obesity and bariatric surgery using their social network platforms (See addendum A). Patients who are interested in participation will be invited to contact the study coordinator. Patients who complete the pre-screening assessment and remain eligible will invited to a screening visit.

Patients who remain eligible to partake will receive further information regarding the study procedures and will be provided with instructions and food items and utensils needed for the first 3-day metabolic experiment. Patients will also be provided with a multivitamin-mineral supplement suitable for patients following bariatric surgery to consume for the duration of the study. Habitual dietary intake will be self-reported using a 3-day food diary. For patients who do not meet all inclusion criteria, any newly identified raised blood glucose, blood pressure, abnormal liver function or decreased kidney function will be reported to the patient and their general practitioner.

The study day will be repeated 7 times, each at a different intake level. The subjects will randomly receive one of seven protein intakes levels during each IAAO experiment (figure 1.). Simple randomization will be conducted using RedCap and allocation tables created in R to allocate a different protein level during each of the visits. Allocation will be concealed from participants. One investigator will be unblinded to allocation as he needs to calculate and physically prepare the study diets based on the specific protein intake level of the given study day. This will not interject bias as the study outcomes are metabolic processes measured by objective biochemical analysis.

Adaptation days protocol Patients will be contacted, and experimental visits scheduled. The study protocol is based on the established IAAO method(26). On two adaptation days prior to the IAAO testing day, patient will consume a maintenance diet providing ad libitum energy intake and protein intake of at 1.5 g/kg ideal body weight. This amount of protein meets current upper-limit of protein requirements for individuals after bariatric surgery(16), and thereby to avoid a catabolic state during the adaptation period.

The maintenance diet will be the participants habitual food intake with the additional of additional protein supplements as necessary. Participants will be allowed to consume one cup of coffee or tea and additional water as needed. Food intake during the 2 days will be recorded to measure protein and energy intake.

Metabolic study days On the study days, patients will visit the ACRONIM study unit at UZ Leuven. Patients will be instructed to arrive for the study visit after a 12-hour fast overnight. On arrival, body weight and body composition will be measured as described above. Patient will receive eight hourly isocaloric meals, each providing 1/12 of their daily energy requirement, thus 67% of their total daily intake.

The 7 test protein intake levels will be testes. It is important that there are at least 2 intake levels below and above the measured protein requirements to identify a breakpoint of amino acid oxidation . Therefore, we selected a range of intake levels which includes two intakes below requirements in healthy men and women, one which is aligned to healthy requirements, and four at higher levels, anticipating that the breakpoint will occur before the final two intake levels.

The remainder of the diet will be provided as 40% fat and 40% carbohydrate to meet daily energy requirements of REE x 1.5. Protein is provided as a crystalline amino acid mixture with a similar amino acid profile to egg protein. The remainder of the diet will be made up of protein-free powder, flavouring, oil, and protein-free cookies.

From the 5th meal the tracer protocol will commence. A primer dosage of 0.176 mg/kg NaH13CO3 and 1.86 mg/kg 1-13C phenylalanine will be provided with the fifth meal. With the next three meals, 1.2 mg/kg 1-13C phenylalanine will be added.

The phenylalanine tracer will form part of a total dietary phenylalanine intake if 30.5 mg/kg/day, approximately three times the Recommended Daily Allowance (RDA,) to ensure sufficient supply for protein synthesis. The RDA for an amino acid is the amount of the amino acid required for protein synthesis, as previously determined by IAAO studies. Equally total tyrosine intake will be 40 mg/kg/day, well in excess of requirements, to minimize the conversion of phenylalanine to tyrosine for protein deposition. Both stable isotopes will be purchased from Cambridge Isotope Laboratories (Woburn, MA, USA).

Breath and urine samples will be collected to measure phenylalanine oxidation and phenylalanine flux respectively. 3 x12ml breath samples will be collected at three time-points and 15ml urine samples at 2 time points prior to commencing the tracer protocol. From 2.5 hours after the start of the tracer protocol until the end of the experiment (hour eight). Breath samples will be collected 6 times (12ml x 3 each time) and urine two times (15ml each time). Breath samples will be stored at room temperature and urine samples will be frozen and stored at -20 ˚C. 13CO2 enrichment of expired air and Urine 13C phenylalanine enrichment will be measured with the use of Gas Chromatography-Mass Spectrometry (GC-MS).

Whole-body phenylalanine flux during isotopic steady state will be calculated according to the model of Matthews et al. as was previously described for IAAO studies. Phenylalanine flux is measured as the dilution of ingested labelled phenylalanine, measured as 13C- phenylalanine in urine. The rate of appearance of 13CO2 in expired air (F13CO2) represents the oxidation of ingested phenylalanine. F13CO2 is calculated according to the model of Matthews et al., using a factor of 0.82 to account of carbon dioxide retained in the bicarbonate pool (32).

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 18 - 65 years,
2. Primary RYGB surgery one to ten years before,
3. Weight stable within 5% over the last 3 months,
4. Normotensive or blood pressure controlled with antihypertensive therapy,
5. Provision of informed consent to participate,

Exclusion Criteria:

1. Current diagnosis of cancer or active cancer in the preceding 1 year,
2. Any chronic or acute disease which is known to affect amino acid absorption, metabolism, or requirements,
3. Weight loss after bariatric surgery of less than 40% of excess weight,
4. Weight regain after bariatric surgery greater than 20% of nadir weight,
5. Diabetes mellitus defined as a fasting plasma glucose concentration ≥ 7.0 mmol, or HbA1c less than 6.5%, or medical treatment for diabetes.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for the study will be recruited among the patients of the Obesity Clinic of the University Hospitals Leuven (UZ Leuven Obesity Clinic) or from individuals recruited through patients-groups.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
estimated average protein requirements | Postprandial plateau in amino acid oxidation, after 8 hours of feeding. 49 studies (7 at 7 protein intake levels each) will be conducted over 6 months to determine to outcome collectively for all participants.
  Estimated protien requirements will be calculated for the total study population, not per participant, and expressed as g/kg bodyweight and g/kg fat free mass

CONTACTS AND LOCATIONS:
Overall Officials: Bart Van der Schueren, MD PhD, Principal Investigator — KU Leuven
Locations (1):
- Universitaire Ziekenhuizen KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Study data will be uploaded to a KU Leuven data repository (RDR) and be made available on request
Time Frame: Study data will be made available upon publication of the results
Access Criteria: Study investigators. Other requests should be directed to the investigators.